CLINICAL TRIAL: NCT03826121
Title: A 12 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Sesame Oil Cake Extract on Improvement of Cognitive Function
Brief Title: Efficacy and Safety of Sesame Oil Cake Extract on Improvement of Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Young Chul Chung, Professor of Psychiatry, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KH_CF_SE
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Cognitive Function
Keywords: Cognitive Function; Sesam Esamesame Oil Cake

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sesame Oil Cake Extract (Experimental): Sesame Oil Cake Extract 1.5 g/day for 12 weeks
  Interventions: Dietary Supplement: Sesame Oil Cake Extract
- Placebo (Placebo Comparator): placebo for 12 weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Sesame Oil Cake Extract — Sesame Oil Cake Extract 1.5 g/day for 12 weeks.
  Arms: Sesame Oil Cake Extract
Dietary Supplement: placebo — placebo for 12 weeks.
  Arms: Placebo

SUMMARY:
This study was the efficacy and safety of Sesame oil cake extract on improvement of Cognitive Function

DETAILED DESCRIPTION:
This study was a 12 weeks, randomized, double-blind, placebo-controlled human trial to evaluate. 70 subjects were participated in Sesame Oil Cake Extract or placebo group. To evaluate the changes of the evaluation items when Sesame Oil Cake Extract was taken three times a day compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Those who are at least 60 years of age at screening
* Those who word list memory / recollection/ recognition test scores of CERAD -K decrease 1-2 SD number of normal value
* Those who agree to voluntary participation and to comply with the Notice after fully hearing and understanding the details of this human trial

Exclusion Criteria:

* Those with a past history of treatment with Axis I disorder in SCID(Structured Clinical Interview for DSM-IV) which is a structured clinical interview in the Diagnostic and Statistical Manual of Mental Disorders at Screening or who have been treated within the last 3 years
* Those with alcohol abuse or dependence within the last 3 months
* Those who have clinically significant following severe illness (Epilepsy, mental retardation, brain nervous system diseases, endocrine diseases, blood / malignant tumors, cardiovascular diseases, Crohn's disease, etc.)
* Those who shows the following results in the Laboratory test

  * AST, ALT > 3 times upper limit of normal range
  * Other significant laboratory test opinion
* Those who take any prescription medicines or herbal medicines within 2 weeks before the first ingestion date or take any OTC or vitamin preparations within 1 week
* Those who participate in other human trial within 2 months before the first ingestion
* Those who whole blood donation within 1 months before the first ingestion or Component blood donation within 2 weeks
* Those who is deemed unsuitable for participating in the human trial due to other reasons

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Changes of Visual learning test | 12 weeks
  Visual learning test was measured in baseline and 12 weeks.
Changes of Visual working memory test | 12 weeks
  Visual working memory test was measured in baseline and 12 weeks.
Changes of Verbal learning test | 12 weeks
  Verbal learning test was measured in baseline and 12 weeks.

SECONDARY OUTCOMES:
Changes of the Montreal Cognitive Assessment(MoCA-K) | 12 weeks
  The cognitive function evaluation using the Montreal Cognitive Assessment(MoCA-K) is a total of 8 items, and evaluates cognitive functions such as time / execution power, vocabulary, memory, attention, sentence, abstraction, delayed recall, and orientation.
  Time / execution power's total score is 5 points, vocabulary's total score is 3 points, attention's total score is 3 points, sentence's total score is 3 points, abstraction's total score is 2 points, delayed recall's total score is 5 points, orientation's total score is 6 points. It takes about 10 minutes to complete, and the total score is 30 points and total score make sum score. A score of 23 points or more is regarded as normal. If you have less than 6 years of education, add 1 point.
  It takes about 10 minutes to complete, and the score is 30 points. A score of 23 points or more is regarded as normal. If you have less than 6 years of education, add 1 point.
Changes of beta-amyloid | 12 weeks
  Beta-amyloid(pg/mL) was measured in baseline and 12 weeks.
Changes of Oxidation index(8-OHdG) | 12 weeks
  Oxidation index(8-OHdG)(ng/mL) was measured in baseline and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Young-chul Chung, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Department of Psychiatry, Chonbuk National University Hospital, Jeonju, South Korea